CLINICAL TRIAL: NCT05406050
Title: Pharmacokinetic and Bioequivalence Study of Eldecalcitol Soft Capsule 0.75 ug in Healthy Chinese Subjects Under Fasting and Fed Conditions: A Randomized, Single-center, Single-dose, Open-label, Two-period Crossover Study
Brief Title: Bioequivalence Study of Eldecalcitol Soft Capsule in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Wenzhou Haihe Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ZJHH-Eld
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR (Experimental): Subjects first receive a single-dose of 0.75 μg test eldecalcitol soft capsule (T, produced by Wenzhou Haihe Pharmaceutical Co., Ltd. China) in the first treatment period and to receive the reference (R, produced by Chugai Pharmaceutical Co., Ltd. Japan) in the second treatment period.
  Interventions: Drug: reference eldecalcitol soft capsule; Drug: test eldecalcitol soft capsule
- RT (Experimental): Subjects first receive a single-dose of 0.75 μg reference eldecalcitol soft capsule (R, produced by Chugai Pharmaceutical Co., Ltd. Japan) in the first treatment period and to receive test capsule (T, produced by Wenzhou Haihe Pharmaceutical Co., Ltd. China) in the second treatment period.
  Interventions: Drug: reference eldecalcitol soft capsule; Drug: test eldecalcitol soft capsule

INTERVENTIONS:
Drug: reference eldecalcitol soft capsule — 0.75 μg, produced by Chugai Pharmaceutical Co., Ltd. Japan
Drug: test eldecalcitol soft capsule — 0.75 μg, produced by Wenzhou Haihe Pharmaceutical Co., Ltd. China

SUMMARY:
A single-center, open-label, randomized, two-period, crossover study design of pharmacokinetics and bioavailability in healthy Chinese subjects under fasting conditions.

DETAILED DESCRIPTION:
Eldecalcitol is a novel active vitamin D3,1,25(OH)2D3 derivative for the treatment of osteoporosis, which was first approved in Japanin 2011. With a hydroxy propoxy substituent at the 2βposition of 1,25(OH)2D3, eldecalcitol not only kept the high safety advantage but also showed much stronger effects on bone, such as improving bone metabolism, increasing bone mineral density(BMD) and preventing new vertebral fracture.Here in this study, we have compared the pharmacokinetic and bioequivalent profiles of two eldecalcitol soft capsule formulations at a single dose of 0.75 μg both under fasting and fed condition in healthy Chinese volunteers.

28 subjects participated in the fasting trial were randomly assigned to two groups to receive a single-dose of 0.75 μg reference eldecalcitol soft capsule (R, produced by Chugai Pharmaceutical Co., Ltd. Japan) or test capsule (T, produced by Wenzhou Haihe Pharmaceutical Co., Ltd. China) with about 240 ml warm water in the first treatment period and to receive another formulation in the second treatment period. There was a 21-day wash-out between the two treatment periods. For those participated in the fed trial, it was almost the same, except that 30 subjects had unified breakfast with high fat and high calories 30 minutes before dosing.Blood samples (8ml) for the determination of eldecalcitol were collected pre-dose and at 0.5,1,2,2.5,3,3.5,4,4.5,5,6,8,10,12,15,24,36,48,72,96,120,144, and 168 h post-dose in the fasting trial. And for those participated in the fed trial, blood samples (8ml) were collected pre-dose and at1,2,3,4,5,6,8,10,12, 14,16,24,28,36,48,72,96,120,144,168, and 192 h post-dose.

ELIGIBILITY:
Inclusion Criteria:

* 1)Subjects are able to give the signed ICF before the study, and fully understand the study content, process and possible adverse reactions;
* 2) Subjects are able to complete the study in compliance the study in compliance with the protocol;
* 3)Subjects (including male subjects) agree to adopt effective contraceptive methods and not plan to get pregnant or to donate sperm or ovum from 14 days before screening to 3 months after study completion;
* 4)Healthy male and female subjects above 18 years of age ( inclusive);
* 5)Ssubjects who are at least 50 kg, with a Body Mass Index (BMI)= Weight/Height2 (kg/m2) between 19.0-28.0 kg/m2 (both inclusive);

Exclusion Criteria:

* 1) allergic to two or more substances or to experimental drugs;
* 2) with a significant history of gastrointestinal inflammation/ulcer or other medical history affecting drug absorption or other diseases not appropriate to attend the trial;
* 3) serious disease, major surgery or a history of trauma 3 months before screening;
* 4) use of any medication including herbal medicine or healthcare products containing calcium, magnesium or vitamin D within 14 days before the first dose;
* 5) use of any investigational drug or product within 3 months prior to the first dose;
* 6) smoking more than five cigarettes a day in the last three months, or cannot quit smoking during the study period;
* 7)alcoholics or drug abuser;
* 8)any abnormality with clinical significance of vital signs, physical examination, laboratory examination and electrocardiograph (ECG) examination;
* 9) consumption of any caffeine-containing food or beverage, any beverage or food with abundant xanthine or any grapefruit or grapefruit-containing juices within 48 hours prior to receiving study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Day0-Day30
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | Day0-Day30
  Evaluation of Area under the plasma concentration versus time curve (AUC0-t)
Area under the plasma concentration versus time curve (AUC0-∞) | Day0-Day30
  Evaluation of Area under the plasma concentration versus time curve (AUC0-∞)
Bioequivalence | Day0-Day30
  Analysis of variance (ANOVA) was performed after logarithmic conversion of main pharmacokinetic parameters (Cmax, AUC) to calculate 90% confidence interval of geometric mean ratio of main pharmacokinetic parameters of the two preparations, and equivalence comparison was conducted. The equivalent interval was set to 80.00%~125.00%

SECONDARY OUTCOMES:
Safety | Day0-Day30
  Collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Dr., Principal Investigator — the study director of phase I clinical research center
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China